CLINICAL TRIAL: NCT01457963
Title: Pulmonary Embolism in Mechanically Ventilated Patients Requiring Computed Tomography: Prevalence, Risk Factors and Outcome
Brief Title: Prevalence of Pulmonary Embolism in ICU
Acronym: PEICU
Status: Completed | Type: Observational
Sponsor: University Hospital, Grenoble (Other)
Responsible Party: Sponsor
Other Study IDs: 5891
Record Dates: First submitted 2011-10-20; First posted 2011-10-24 (Estimated); Last update posted 2011-10-24 (Estimated); Status verified 2011-10

CONDITIONS: Pulmonary Embolism; Deep Venous Thrombosis
MeSH Terms: conditions — Pulmonary Embolism; Venous Thrombosis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- pulmonary embolism, deep venous thrombosis

SUMMARY:
The primary objective of this study was to estimate the prevalence of PE among consecutive ICU patients receiving MV who required thoracic computed tomography (CT) with contrast agent injection, regardless of whether PE was suspected clinically. The secondary objectives were to assess the association between PE and DVT, to identify risk factors for VTE, and to determine the outcome of VTE.

DETAILED DESCRIPTION:
Background: Pulmonary embolism (PE) produces nonspecific or minimal symptoms in mechanically ventilated (MV) patients, leading to underdiagnosis. We estimated the prevalence of PE and associations with deep vein thrombosis (DVT) among MV patients.

Methods: Consecutive MV patients who required thoracic computed tomography (CT) in a single ICU. Compression ultrasound of the four limbs was performed within 48 hours of inclusion. Curative anticoagulation therapy was given immediately after PE diagnosis.

ELIGIBILITY:
Inclusion Criteria:

* all patients requiring invasive MV and thoracic contrast-enhanced CT for any reason

Exclusion Criteria:

* a diagnosis of PE before ICU admission,
* allergy to contrast agents,
* and age younger than 18 years.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients in ICU, mecanically ventilated with a CT scab with iodine injection
Sampling Method: Non-Probability Sample
Enrollment: 176 (Actual)
Dates: Start 2009-12; Primary Completion 2011-04 (Actual); Study Completion 2011-04 (Actual)

PRIMARY OUTCOMES:
Find a pulmonary embolism on the CT scan | CT scan at the day of inclusion
  TO estimate the prevalence of PE among consecutive ICU patients receiving MV who required thoracic computed tomography (CT) with contrast agent injection, regardless of whether PE was suspected clinically.

SECONDARY OUTCOMES:
To find thrombus on compression ultrasound (CUS) of the four limbs | CUS within 48 hours after the CT scan

CONTACTS AND LOCATIONS:
Overall Officials: Jean Francois TIMSIT, PU/PH, Principal Investigator — University Hospital, Grenoble
Locations (1):
- University hospital of grenoble, Grenoble, France

REFERENCES:
- [Derived] Minet C, Lugosi M, Savoye PY, Menez C, Ruckly S, Bonadona A, Schwebel C, Hamidfar-Roy R, Dumanoir P, Ara-Somohano C, Ferretti GR, Timsit JF. Pulmonary embolism in mechanically ventilated patients requiring computed tomography: Prevalence, risk factors, and outcome. Crit Care Med. 2012 Dec;40(12):3202-8. doi: 10.1097/CCM.0b013e318265e461. PMID 23164766